CLINICAL TRIAL: NCT07027423
Title: A Phase 1b Trial of BOLD-100 Plus Doxorubicin in Advanced Soft Tissue Sarcomas
Brief Title: BOLD-100 Plus Doxorubicin in Advanced Soft Tissue Sarcomas
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BOLDSARC-01
Record Dates: First submitted 2025-04-30; First posted 2025-06-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Sarcoma, Soft-tissue; Sarcoma; Sarcoma,Soft Tissue; Sarcomas
MeSH Terms: conditions — Sarcoma | interventions — KP 1339; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BOLD-100 and Doxorubicin Dose Level -1 (Experimental): Escalation phase DL-1 - BOLD-100 230mg/m^2 + Doxorubicin
  Interventions: Drug: BOLD-100; Drug: Doxorubicin 75 mg/m^2
- BOLD-100 and Doxorubicin Dose Level 1 (Experimental): Escalation phase DL1 - BOLD-100 420mg/m^2 + Doxorubicin
  Interventions: Drug: BOLD-100; Drug: Doxorubicin 75 mg/m^2
- BOLD-100 and Doxorubicin Dose Level 2 (Experimental): Escalation phase DL2 - BOLD-100 500mg/m^2 + Doxorubicin
  Interventions: Drug: BOLD-100; Drug: Doxorubicin 75 mg/m^2
- BOLD-100 and Doxorubicin Dose Level 3 (Experimental): Escalation phase DL3 - BOLD-100 625mg/m^2 + Doxorubicin
  Interventions: Drug: BOLD-100; Drug: Doxorubicin 75 mg/m^2
- BOLD-100 and Doxorubicin (Experimental): Exapsnion: BOLD-100 (RP2D) and Doxorubicin
  Interventions: Drug: BOLD-100; Drug: Doxorubicin 75 mg/m^2

INTERVENTIONS:
Drug: BOLD-100 — BOLD-100 in combination with Doxorubicin (Escalation)
  Arms: BOLD-100 and Doxorubicin Dose Level -1; BOLD-100 and Doxorubicin Dose Level 1; BOLD-100 and Doxorubicin Dose Level 2; BOLD-100 and Doxorubicin Dose Level 3
Drug: Doxorubicin 75 mg/m^2 — BOLD-100 in combination with Doxorubicin (Escalation)
  Arms: BOLD-100 and Doxorubicin Dose Level -1; BOLD-100 and Doxorubicin Dose Level 1; BOLD-100 and Doxorubicin Dose Level 2; BOLD-100 and Doxorubicin Dose Level 3
Drug: BOLD-100 — BOLD-100 in combination with Doxorubicin (Expansion)
  Arms: BOLD-100 and Doxorubicin
Drug: Doxorubicin 75 mg/m^2 — BOLD-100 in combination with Doxorubicin (Expansion)
  Arms: BOLD-100 and Doxorubicin

SUMMARY:
A Phase 1b, non-randomized, single-institution trial designed to assess the safety, tolerability and the highest dose with acceptable toxicity (RP2D) of BOLD-100 in combination with doxorubicin in patients diagnosed with advanced soft tissue sarcomas. The trial is divided into two phases: an initial dose-escalation phase for BOLD-100, followed by a dose-expansion phase based on the recommended dose for Phase 2. In the dose-escalation phase, we plan to enroll 12-15 patients, with an additional 17 patients in the dose-expansion phase.

Participants will receive BOLD-100 intravenously on Days 1 and 8 of a 21-day cycle, in combination with doxorubicin (75 mg/m², intravenous) administered on Day 1 of each 21-day cycle for up to six cycles. Participants will continue to receive BOLD-100 for as long as the cancer is not getting worse, The maximum cycles of doxorubicin are 6 cycles.

Participants will undergo a screening assessment prior to the start treatment to determine eligibility for enrollment. Treatment will commence on Day 1 and will continue until the protocol-defined criteria for treatment withdrawal are met. Disease response will be assessed using CT or MRI scans, starting at 12 weeks after the initiation of treatment and continuing every 12 weeks until withdrawal.

Upon treatment discontinuation or study withdrawal, a post-treatment assessment will be conducted at end of treatment and at 30 days of the last BOLD-100 dose, with follow-up visits scheduled every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent in accordance with federal, local, and institutional guidelines.
2. Age > 18 years.
3. Patients must have histologically confirmed locally advanced/unresectable or metastatic soft tissue sarcoma of limited subtype LMS, DDLPS and UPS (including Myxofibrosarcoma-MFS).
4. Patients be systemic treatment naïve, with incurable, advanced or metastatic disease.
5. Patient must have measurable disease as defined by RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate hematopoietic function:

   1. total white blood cell (WBC) count ≥2000/mm3.
   2. absolute neutrophil count (ANC) ≥1500/mm3.
   3. platelet count ≥100,000/mm3.
8. Adequate hepatic function:

   1. Bilirubin <2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN).
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 X ULN. In the case of known (radiological and/or biopsy documented) liver metastasis, ALT/AST <5.0 X ULN is acceptable.
9. Adequate renal function defined as <1.5x upper limits of normal
10. Cardiac function: A normal left ventricular ejection fraction (LVEF) of > 50% as evidenced by an echocardiogram or nuclear medicine study performed within 28 days of the proposed study commencement.
11. Female patients of childbearing potential must agree to use two methods of contraception (including one highly effective and one effective method of contraception) and have a negative serum pregnancy test at 72 hours prior to receiving the first dose of study medication. Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Patient is pregnant or lactating.
2. Radiation (except planned or ongoing palliative radiation outside of the region of measurable disease), chemotherapy, immunotherapy, any other systemic anticancer therapy, or participation in an investigational anti-cancer study ≤3 weeks prior to initiation of therapy.
3. Major surgery within 4 weeks before initiation of therapy.
4. Prior systemic therapy.
5. Unstable cardiovascular function:

   1. symptomatic ischemia, or.
   2. uncontrolled clinically significant conduction abnormalities (e.g., ventricular tachycardia on anti-arrhythmic is excluded and 1st degree AV block or asymptomatic LAFB/RBBB will not be excluded) or.
   3. congestive heart failure (CHF) of NYHA Class ≥3, or.
   4. myocardial infarction (MI) within 3 months of initiation of therapy.
6. Active, ongoing or uncontrolled active infection within one week prior to first dose.
7. Malignancies other than disease under study within 2 years prior to Cycle 1, Day 1, except for those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ). Prior chemotherapy is allowed apart from regimens that contained anthracycline based therapies.
8. Known to be HIV seropositive.
9. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or hepatitis B virus (HBV) surface antigen (HBsAg).
10. Patients with active CNS malignancy. Asymptomatic small lesions are not considered active. Treated lesions may be considered inactive if they are stable for at least 3 months.
11. Serious psychiatric or medical conditions that could interfere with treatment.
12. Concurrent therapy with approved or investigational anticancer therapeutic agents.
13. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicities (DLTs) | Entire duration of Cycle 1 (21 day cycle)
The rate of Adverse Events (AE) | time the consent form is signed through 12 months following cessation of treatment
  The rate of Adverse Events (AE) characterized by type, frequency, severity graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0
Rate of toxicities | time the consent form is signed through 12 months following cessation of treatment.
  Rate of toxicities as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0, adverse events (AEs), serious AEs (SAEs), dose interruptions and assessment.
Participant Quality of Life | pre-dose, Cycle 2 Day1, Cycle 7 Day 1, Cycle 12 Day 1 (21 day cycles)
  Assessed using EORTC QLQ-C30 (European Organization For Research And Treatment Of Cancer, Core Quality of Life Questionnaire). With scores from 0 to 100. A high scale score represents a higher response level.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | time the consent form is signed through treatment completion, up to 4-6 weeks after progression if applicable
  Progression-free survival (PFS), response rate using RECIST v 1.1, clinical benefit rate (CR, PR, SD >16 weeks) using the Kaplan Meier method to estimate with corresponding 95% CI
Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 | During Cycle 1 pre-dose, 1hour, 2hours and 48hours post-dose, through Cycle 2 pre-dose (21 day cycles)
  Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 (in the first 3 patients per dose level) using Peak Plasma Concentration (Cmax), which will be compared to single agent population PK of doxorubicin and BOLD-100.
Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 | During Cycle 1 pre-dose, 1hour, 2hours and 48hours post-dose, through Cycle 2 pre-dose (21 day cycles)
  Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 (in the first 3 patients per dose level) using area under the plasma concentration versus time curve (AUC), which will be compared to single agent population PK of doxorubicin and BOLD-100.
Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 | During Cycle 1 pre-dose, 1hour, 2hours and 48hours post-dose, through Cycle 2 pre-dose (21 day cycles)
  Analysis of pharmacokinetic parameters of doxorubicin and BOLD-100 (in the first 3 patients per dose level) using time to peak drug concentration (Tmax), which will be compared to single agent population PK of doxorubicin and BOLD-100.

OTHER OUTCOMES:
Correlate cellular morphology and biomarker changes | through study completion, an average of 1 year
  Correlate cellular morphology and biomarker changes on sarcoma biopsy specimens compared to archival tissue. Immunohistochemical expression/localization of GRP78.
Correlate immune signatures and expression of GRP78 levels | through study completion, an average of 1 year
  Correlate immune signatures and expression of GRP78 levels in leukocytes in patients' blood with response rate using non-parametric Wilcoxon rank sum.

CONTACTS AND LOCATIONS:
Locations (1):
- UHN- Princess Margaret Cancer Center, Toronto, Ontario, Canada